CLINICAL TRIAL: NCT06717438
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Study of Zatolmilast (BPN14770) in Subjects With PPP2R5D Neurodevelopmental Disorder (Jordan's Syndrome)
Brief Title: Study of Zatolmilast (BPN14770) in Participants With PPP2R5D Neurodevelopmental Disorder (Jordan's Syndrome [JS])
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPN14770-CNS-205
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Jordan's Syndrome; PPP2R5D Neurodevelopmental Disorder
Keywords: Jordan's Syndrome; JS; PPP2R5D Neurodevelopmental Disorder; Zatolmilast; BPN14770
MeSH Terms: interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPN14770 (Experimental): Participants will receive a weight adjusted dose of BPN14770 twice daily (BID) during the 24-week Double-blind Period.
  Participants in the BPN14770 arm who complete the Double-blind Period will have the opportunity to continue in the Open-label Extension Period. Participants will receive a weight adjusted dose of BPN14770 BID during the 24-week Open-label Extension Period.
  Interventions: Drug: BPN14770
- Placebo (Placebo Comparator): Participants will receive BPN14770 matching placebo BID during the 24-week Double-blind Period.
  Participants in the placebo arm who complete the Double-blind Period will have the opportunity to continue in the Open-label Extension Period. Participants will receive a weight adjusted dose of BPN14770 BID during the 24-week Open-label Extension Period.
  Interventions: Drug: BPN14770; Drug: Placebo

INTERVENTIONS:
Drug: BPN14770 — Capsules for oral administration
  Other Names: Zatolmilast
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of BPN14770 in participants aged 9 to 45 years with JS.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 9 to 45 years, inclusive.
2. Participant has confirmed/documented history of PPP2R5D Neurodevelopmental Disorder.
3. Current treatment with no more than 3 prescribed psychotropic medications.
4. Participant has a parent, legal authorized guardian or consistent caregiver.

Exclusion Criteria:

1. Participant has body weight less than 25 kilograms (kg).
2. Clinically significant abnormalities, in the investigator's judgment, in safety laboratory tests, vital signs, or electrocardiogram (ECG), as measured during Screening.
3. Concurrent major psychiatric condition (e.g., Major Depressive Disorder, Schizophrenia or Bipolar Disorder) as diagnosed by the investigator. Participants with additional diagnosis of Autism Spectrum Disorder or Anxiety Disorder will be allowed.
4. Participant is planning to commence psychotherapy or cognitive behavior therapy (CBT) during the period of the study or had begun psychotherapy or CBT within 4 weeks prior to Screening.

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Week 50
Discontinuation-emergent Signs and Symptoms (DESS) Questionnaire Score | Week 50
Number of Participants with Seizures | Up to Week 50
Number of Participants at Suicidality Risk | Up to Week 48

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No